CLINICAL TRIAL: NCT00077038
Title: Modulation of the Visual Information Processing in the Human Parieto-Frontal Network as Studied by a Frequency Tagging Technique During Visuomotor Tracking
Brief Title: Brain Activity in Visual-Motor Behavior
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040117; 04-N-0117
Record Dates: First submitted 2004-02-09; First posted 2004-02-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Healthy
Keywords: Visual Feedback; Cortical Connectivity; Magnetoencephalography; Eye Tracking; Healthy Volunteer; HV

SUMMARY:
This study will examine how the brain works when people look at an object, follow a moving object with their eyes, and reach out their hand to an object. Different areas of the brain work together in reaching out a hand to an object. These areas are also important for concentrating on objects or following them with the eyes. This study will use magnetoencephalography (MEG) to observe more precisely how discrete parts of the brain work during these movements. MEG is a new technique for recording magnetic field changes produced by brain activity.

Healthy normal volunteers 20 years of age and older who are right-handed and who have no history of brain or eye disease may be eligible for this study. Candidates will be screened with a medical history and brief physical examination. They will complete questionnaires for MEG screening and for determining handedness.

Participants undergo MEG recording and magnetic resonance imaging (MRI). For MEG, the subject sits comfortably in front of a computer screen, and a cone containing magnetic field detectors is lowered onto the head. Electrodes are placed on both sides of the outer part of the eyelids and just above and below the left eye to monitor eye movement. During MEG, subjects perform the following tasks:

1. Eye fixation: A small white cross and a white ring appear on the center of the computer screen. Another white ring moves slowly around the screen in random fashion. Subjects keep their eyes fixed on the central cross and concentrate on the ring at the center, ignoring the moving ring.
2. Ocular tracking: The same cross and rings in task 1 appear on the screen, but in this task the subjects follow the moving ring with their eyes and ignore the cross and ring in the center.
3. Peripheral manual tracking task (right hand): In addition to the cross and rings in task 1, a small white disc-shaped cursor appears on the screen. Using their right hand, subjects use a joystick to move the cursor as precisely as possible to follow the moving ring, while keeping their eyes fixed on the central cross.
4. Peripheral manual tracking task (left hand): The same as task 3, except using the left hand.
5. Central manual tracking: The cross, rings, and joystick are the same as in task 3. Subjects move the cursor to follow the moving ring as precisely as possible, while following the moving ring with their eyes and ignoring the cross and ring in the center of the screen.

Subjects practice each task before MEG recording starts. Then they perform each task twice in random order, with a 1- or 2-minute break between tasks.

Subjects who do not have previous MRI images filed in NINDS's database undergo MRI scanning. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The scanner is a metal cylinder surrounded by a strong magnetic field. Subjects lie still on a table that can slide in an out of the cylinder. They can communicate with the MRI staff at all times during the procedure.

DETAILED DESCRIPTION:
HYPOTHESIS:

The hypothesis of this study is that the parieto-frontal network is activated by visuomotor behavior in humans.

OBJECTIVES:

To detect frontal and parietal cortical activity during a visuomotor task with frequency modulated visual stimuli using magnetoencephalography (MEG).

To reveal how the parieto-frontal activities change according to different conditions of attention, gaze, and motor output.

STUDY POPULATION:

Right handed normal volunteers with no known history of neurological or ophthalmological diseases will be recruited to participate in this study.

DESIGN:

This study is a combination of a frequency tagging method and an MEG. Visual stimuli are presented, flickering in specific (tagged) frequencies. The cortical distribution of the visual information is estimated from the tagged frequency response of the MEG signal. We will use a visuomotor tracking task with a multifactorial task design (attention, target motion, position in retinal coordinate, and manual tracking) to evaluate the effect of each factor separately.

OUTCOME MEASURES:

We will use the adaptive linear-filter technique known as synthetic aperture magnetometry (SAM) to estimate the source location and strength of the tagged frequencies. The estimated cortical source activity power at the frontal and parietal cortices will be group analyzed with multiple logistic models and by analysis of variance (ANOVA) with correction for multiple comparisons.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects must be 20 years old or older and right-handed as screened by Edinburgh handedness inventory.

They must be healthy and have no known history of neurological or ophthalmological diseases.

EXCLUSION CRITERIA:

Subjects under the age of 20 will be excluded from this study.

Subjects who match the criteria below will be excluded from this study due to human subject protection and because they may negatively affect the MEG data quality.

Subjects wearing glasses.

Subjects with involuntary movement or dyskinesia.

Subjects with spontaneous nystagmus.

Subjects who can not execute the eye or manual tracking after sufficient practice time.

Subjects with metal objects in the body.

Subjects with history of severe head trauma.

Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-02-06; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Glover S. Optic ataxia as a deficit specific to the on-line control of actions. Neurosci Biobehav Rev. 2003 Aug;27(5):447-56. doi: 10.1016/s0149-7634(03)00072-1. PMID 14505686